CLINICAL TRIAL: NCT02231801
Title: Vital Sign Monitoring of Mother-Infant Dyads During Kangaroo Care in Preterm Infants
Brief Title: Monitoring of Vital Signs During Skin-to-skin Holding by Mothers of Their Preterm Babies
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 14-1323; PD14-03941
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Other Preterm Infants
Keywords: Preterm; Kangaroo Care; Skin-to-Skin; Vital Sign; Heart Rate; Respiratory Rate; Oxygen Saturation
MeSH Terms: conditions — Premature Birth | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mother-Infant Dyad: Skin-to-skin holding of preterm infants by their mothers
  Interventions: Behavioral: Mother-Infant Dyad

INTERVENTIONS:
Behavioral: Mother-Infant Dyad — Skin-to-skin holding of preterm infants by their mothers
  Other Names: Kangaroo Care

SUMMARY:
This observational study aims to monitor the vital sign changes in both mother and baby that occur during kangaroo care in preterm infants and to investigate any potential correlations between maternal measurement values and those of the infant. The purpose of this observational study is to look for a method to track the earliest responses that could, theoretically, be considered as 'social responses' in hopes of providing developmental interventions earlier to at-risk infants.

DETAILED DESCRIPTION:
The goal of this observational study is to identify any signs of early "social response" in order to be able to assist infants that lack this response with early neurobehavioral modifications.

ELIGIBILITY:
Inclusion Criteria:

* inborn at Mount Sinai
* gestational age between 30 0/7 weeks and 34 6/7 weeks gestation
* only one infant of a multiple gestation
* plan by family to do kangaroo care during NICU stay

Exclusion Criteria:

* outborn infants
* gestational age less that 29 6/7 weeks or greater than 35 0/7 weeks
* other infants of multiple gestation (see inclusion criteria)
* any major congenital anomalies
* sepsis and/or any other serious clinical complication precluding kangaroo care

Ages: 30 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born at Mt. Sinai Hospital and admitted to the NICU. Preterm infants between 30 0/7 weeks gestational age to 34 6/7 weeks gestation age.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Heart Rate | up to 30 minutes

SECONDARY OUTCOMES:
Respiratory Rate | up to 30 minutes
Oxygen Saturation | up to 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ian Holzman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States